CLINICAL TRIAL: NCT07073222
Title: Development and Evaluation of an Escape Room for Nursing Students Taking Pharmacology Course
Brief Title: An Escape Room for Nursing Students Taking Pharmacology Classes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Nurhan Aktaş, assistant professor, Kahramanmaraş İstiklal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Istiklal University
Record Dates: First submitted 2025-06-29; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Nursing Student; Pharmacology
Keywords: escape room; pharmacology; gamification; nursing students

STUDY DESIGN:
Masking Description: There is nothing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Escape room playgroup (Experimental): Escape room game is played with escape room game group
  Interventions: Other: Escape room game

INTERVENTIONS:
Other: Escape room game — Escape room games are live action team-based games where players discover clues, solve puzzles and complete tasks in one or more rooms to accomplish a specific goal within a limited time.

SUMMARY:
The study was planned as a pre-test-post-test single-group, quasi-experimental design to evaluate the effects of the education provided with the escape room game on the level of autonomic nervous system drug knowledge and perceptions of the game experience in nursing students taking the Pharmacology course. The sample of the study will consist of students enrolled in the Nursing Pharmacology course at the Kahramanmaraş İstiklal University, Faculty of Health Sciences, Department of Nursing in the 2024-2025 academic year, who meet the research criteria and agree to participate in the study. The study will be conducted in two stages. In the first stage, the necessary materials for the game development and evaluation process will be prepared and the content validity study of these materials will be conducted. In the second stage, the escape room game will be applied and data will be collected. The data will be collected with the "Descriptive Characteristics Form" and the "Autonomic Nervous System Drug Knowledge Test" (pre-test) before the escape room game, and with the "Autonomic Nervous System Drug Knowledge Test" (post-test) and the "Game Playing Experience Scale" after the game. The analysis of the data will be completed by transferring it to the IBM SPSS Statistics 23 program.

H1a = There is a difference between the mean scores of the autonomic nervous system knowledge test of the students who participated in the escape room game before and after the game.

H1b = There is no difference between the mean scores of the autonomic nervous system knowledge test of the students who participated in the escape room game before and after the game

DETAILED DESCRIPTION:
The research was planned in a pretest-posttest one-group, quasi-experimental design design in order to evaluate the effect of the training given with the escape room game on the autonomic nervous system drug knowledge level of the students and their perceptions of the game experience in nursing students taking the Pharmacology course. The population of the study will consist of students enrolled in the Pharmacology Course for Nurses at Kahramanmaraş İstiklal University, Faculty of Health Sciences, Department of Nursing in the 2024-2025 academic year. In the research, it is planned to reach the universe and no sampling calculation was made. The sample of the research will consist of the students enrolled in the Pharmacology Course for Nurses at Kahramanmaraş İstiklal University, Faculty of Health Sciences, Department of Nursing in the 2024-2025 academic year, who meet the research criteria and who agree to participate in the research. The research will be conducted in two stages. In the first stage, the materials required for the game development and evaluation process will be prepared and the content validity study of these materials will be carried out. In the second stage, the escape room game will be applied and the data will be collected. The data will be collected before the escape room game with "Descriptive Characteristics Form" and "Autonomic Nervous System Drug Knowledge Test" (pre-test), and after the game with "Autonomic Nervous System Drug Knowledge Test" (post-test) and "Game Playing Experience Scale". Data analysis will be completed by transferring to IBM SPSS Statistics 23 programme. Frequency distribution (number, percentage) for categorical variables and descriptive statistics (mean, standard deviation, minimum, maximum) for numerical variables will be given. Parametric and nonparametric tests will be used according to the normal distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* First time registration in Pharmacology Course for Nurses,
* Volunteering to participate in the research

Exclusion Criteria:

* Having a high school, associate degree or bachelor's degree in a health-related field,
* Having difficulty in understanding and speaking Turkish.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Autonomic Nervous System Pharmacology Knowledge Level | Before starting the escape game
  Autonomic Nervous System Pharmacology Knowledge Test (ANSPKT) measures the knowledge level of the study participants.
  ANSPKT contains 20 five-option multiple-choice questions (a minimum score of 0 and a maximum score of 20) on autonomic nervous system pharmacology, including sympathetic nervous system drugs (5 questions), parasympathetic nervous system drugs (5 questions), the effects of the autonomic nervous system on the body (5 questions), and autonomic nervous system neurotransmitters and receptors (5 questions). This test was evaluated by 40 second-year nursing students. Item analysis was conducted to calculate item difficulty and discrimination. Additionally, the test's KR20 reliability criterion was examined. According to the item analysis, the test was found to be of medium difficulty (0.65) and the KR-20 was found to be 0.76, indicating reliability.

SECONDARY OUTCOMES:
Autonomic Nervous System Pharmacology Knowledge Level | ANSPKT was applied to the participants one week after the escape room game.
  After the escape room game, the knowledge level of the participants is evaluated with the Autonomic Nervous System Pharmacology Knowledge Test (ANSPKT).
  The ANSPKT consists of 20 five-option multiple-choice questions (the lowest possible score is 0, and the highest is 20) related to autonomic nervous system pharmacology, including sympathetic nervous system drugs (5 questions), parasympathetic nervous system drugs (5 questions), the effects of the autonomic nervous system on the body (5 questions), and autonomic nervous system neurotransmitters and receptors (5 questions). This test was evaluated by 40 second-year nursing students. The ANSPKT item analysis was conducted to calculate item difficulty and item discrimination values. Additionally, the test's KR20 reliability measure was examined. According to the item analysis results, the test was found to be of medium difficulty (0.65) and the KR-20 was found to be 0.76, indicating that the test was reliable.
perception of game experience | a week after the escape room game
  After the escape room game, participants' game experience perceptions are evaluated with the Gameful Experience Scale (GAMEX).
  GAMEX was developed by Eppman et al. (2018) to assess participants' gaming experience. A Turkish validity and reliability study was conducted with nursing students by Çömez İkican et al. (2024). The scale consists of a total of 27 items and 5 subdimensions. The subdimensions are enjoyment, immersion in the game, creative thinking and emotional activation, absence of negative effects, and mastery. A 5-point Likert-type scale is used in the evaluation of the scale, with scores of "Never" (1), "Rarely" (2), "Sometimes" (3), "Frequently" (4), and "Always" (5). Items 18, 21, 22, and 23 of the scale are scored reversely ("Never" (5), "Rarely" (4), "Sometimes" (3), "Frequently" (2), and "Always" (1). In the original and validity-reliability study of the scale, the Cronbach alpha value for the entire scale was found to be 0.89.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Istiklal University, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No